CLINICAL TRIAL: NCT00693797
Title: Clinical Significance of Collagen Metabolism Changes in Patients With Failing and Pressure Overloaded Left Cardiac Ventricle.
Brief Title: Clinical Significance of Collagen Metabolism Changes in Left Cardiac Ventricle
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government)
Responsible Party: M.Zeman, Faculty hospital, Královské Vinohrady, Prague , Czech Republic
Other Study IDs: NR/9022-3
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Aortic Stenosis
Keywords: ventricular hypertrophy; collagen; aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — frozen serum for collagen metabolism detection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- I, observation: patients with aortic stenosis
- II, observation: patients with aortic stenosis

SUMMARY:
As there are no clinical data in cardiology about the relationship between metabolism collagen changes and their clinical significance, the investigators will check the hypothesis that collagen metabolism changes, detected by biochemical markers for collagen metabolism, could predict the left ventricle remodelling and prognosis in patient with clinically significant pressure overloaded left ventricle.

DETAILED DESCRIPTION:
Clinical assessment and endpoints:

1ST day (the day of entering the hospital or the day of the first contact): Informed consent (see below), clinical examination, ECG, complete echocardiography evaluating the function of the left ventricle (EF) and the presence and the significance of valvular disease, basic laboratory tests incl. CKMB, troponin I, taking of blood samples (5 ml) for the detection of collagen metabolism markers serum level, X-ray of chest, 2nd-3rd day: clinical examination, ECG, basic laboratory tests incl.CKMB, troponin I (only group I) 4th day: clinical check up, ECG, echocardiography, taking of blood samples (5ml) for the detection of collagen metabolism markers serum level (only group I) 30th day: clinical examination l, ECG, echocardiography, taking of blood samples (5ml) for the detection of collagen metabolism markers serum level, 24 hrs ECG monitoring (holter) 6 months: clinical examination, ECG, echocardiography, taking of blood samples (5ml) for the detection of collagen metabolism markers serum level, holter monitoring

1 year: history, clinical examination

Primary endpoint: combined clinical endpoint: death/repeated hospitalisation due to heart failure/myocardial infarction within 30 days and during 1 year follow up.

Secondary endpoints: rehospitalisation for cardiovascular reason, clinically significant arrhythmias, correlations between left ventricle parameters evaluated by echocardiography and collagen metabolism changes evaluated by serum markers

ELIGIBILITY:
Inclusion Criteria:

1. isolated severe aortic stenosis (index aortic valve area less than 0,5 cm2/m2 or mean transaortic pressure gradient more than 40 mm Hg, assessed by echocardiography) and left ventricular hypertrophy (see above)
2. signed informed consent

Exclusion Criteria:

1. presence of more than mild aortic regurgitation or other significant valvular lesion
2. impossibility to obtain echocardiographic tracing of good quality
3. all other diseases, which significantly influence collagen metabolism (renal failure, insulin dependent diabetes mellitus, bone diseases, hepatic failure)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with aortic stenosis and left ventricular hypertrophy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome: combined clinical endpoint: death/repeated hospitalisation due to heart failure/myocardial infarction within 30 days and during 1 year follow up. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jirmář Radovan, M.D., Ph.D., Principal Investigator — Faculty hospital Královské Vinohrady
Locations (1):
- Faculty hospital Královské Vinohrady, Prague, Czechia